CLINICAL TRIAL: NCT00580372
Title: Phase II Study of Intensive "TOTAL THERAPY" for Untreated or Minimally Treated Patients With Multiple Myeloma
Brief Title: UARK 89-001 Phase II Study of Intensive "TOTAL THERAPY" For Untreated or Minimally Treated Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01332
Record Dates: First submitted 2007-12-18; First posted 2007-12-24 (Estimated); Results first posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Treatment (Experimental): Protocol therapy consists of a remission induction phase with mutually non-cross resistant combinations of vincristine, adriamycin, dexamethasone (VAD), high-dose cyclophosphamide with stem cell procurement and etoposide, dexamethasone, cytarabine, cisplatin (EDAP) followed by two courses of melphalan-based high-dose therapy supported by autologous stem cell transplants 4-6 months apart. Maintenance with interferon alpha will be administered until disease progression.
  Interventions: Drug: VAD; Drug: High-Dose cyclophosphamide; Procedure: Hemopoietic stem cell procurement; Drug: EDAP; Procedure: Autologous Hemopoietic Stem Cell Transplant 1; Procedure: Autologous Hemopoietic Stem Cell Transplant 2; Drug: Maintenance

INTERVENTIONS:
Drug: VAD — 3 Cycles (3rd cycle optional): Vincristine 0.5 mg/d d 1 - 4 CI Adriamycin 10 mg/m2/d d 1 - 4 CI Dexamethasone 40 mg/d d 1-4, 9-12, 17-20
Drug: High-Dose cyclophosphamide — Approximately 5-6 weeks after VAD 2 or 3:
  Cytoxan 1.2g/m2/d d 1 - 5 Mesna 3.6 g/m2 d 1
Procedure: Hemopoietic stem cell procurement — Collection target = 10 x 10^6 cells/kg
Drug: EDAP — Approximately 5-6 weeks after high-dose cyclophosphamide Etoposide 100 mg/m2/d d 1 - 4 CI Cisplatin 25 mg/m2/d d 1 - 4 CI Ara C l g/m2 d 5 Dexamethasone 40 mg d 1-5
Procedure: Autologous Hemopoietic Stem Cell Transplant 1 — 4-6 weeks after EDAP: Melphalan 100 mg/m2 days -1 and -2
Procedure: Autologous Hemopoietic Stem Cell Transplant 2 — 4-6 months after Transplant 1: Melphalan 100 mg/m2 days -1 and -2
Drug: Maintenance — 3 months after Transplant 2: Intron A 3 X 10^6 units /m2 M-W-F subcutaneously until relapse

SUMMARY:
This experimental study evaluates the effects of a series of intensive drug regimens as initial treatment for Multiple Myeloma followed by 2 bone marrow transplantations 4-6 months apart in support of high-dose Melphalan, followed by Interferon treatment indefinitely.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated patients with the diagnosis of multiple myeloma are eligible. Similarly, patients who have not had more than one cycle of standard chemotherapy or up to one month of interferon and/or glucocorticoids are eligible.
* Patients must have objective evidence of, or be symptomatic from, complications due to myeloma (e.g., bone pain from fractures, weakness from anemia). Asymptomatic patients may be treated only if the diagnosis is confirmed and if there is evidence of increasing tumor mass (e.g., rising myeloma protein and/or increasing lytic lesions).
* Asymptomatic patients with idiopathic monoclonal peaks, localized plasmacytomas, or indolent, asymptomatic myeloma are not eligible for this study. Any patient without documented increasing disease and/or clearly symptomatic disease is not eligible.
* Measurable, direct manifestations of myeloma must be present, such as monoclonal serum or urine globulins. Plasma cell tumors must also be documented. Patients without protein criteria are eligible if bone marrow has > 30% plasmacytosis documented by bilateral bone marrow aspirations and biopsies.
* Patients with all stages of multiple myeloma (I, II, III) are eligible. Necessary baseline studies must be obtained to determine the stage prior to registration.
* Patients may have received local radiation to painful compression fractures or lytic bone lesions, provided that adequate autologous bone marrow can still be harvested. Patients presenting with clinical conditions requiring radiotherapy (e.g. spinal cord compression) may proceed with concurrent local radiation and VAD. Should compression fractures of known prestudy lytic lesions occur during later, more myelosuppressive phases of induction therapy, radiotherapy should be completed first prior to proceeding with high-dose cyclophosphamide, EDAP or melphalan.
* Patients should be older than 15 years of age and may be up to 65 years old.
* Pregnant females are excluded from study.
* Eligibility criteria change with the progress through the different phases of the induction program towards the two cycles of marrow-ablative therapy. These are summarized in the eligibility checklist.
* Briefly, prior to VAD, patients must have a normal cardiac ejection fraction of > 50% (on ECHO cardiography or MUGGA scan), and fairly normal liver function tests (bilirubin < 2 mg% and serum transaminase levels less than 2 x normal). Screening for viral hepatitis should be negative for acute or chronic active hepatitis. Positive antibody (anti-HAV, HBSAb) suggestive of remote exposure is acceptable. However, patients who test positive for Hepatitis C antibody (anti-HCV) or HIV are ineligible. Those with renal failure are eligible and should start VAD promptly and receive additional medical measures as needed. Patients presenting with infections upon presentation shall receive proper medical management prior to starting therapy. Patient's performance status is not a criterion for entry on the VAD portion of this program.
* After 2 or 3 cycles of VAD, serum creatinine levels must be 2 mg% and carbon monoxide diffusion capacity 50%. Cardiac and liver function requirements as with VAD.
* Not until reaching the high-dose melphalan stage of 70 mg/M2 will there be a requirement for Zubrod performance of 0 and 1 which must also be fulfilled with each of the 2 marrow-ablative doses of melphalan (200 mg/M2).

Exclusion Criteria:

* Less than 10 x 108 cells/kg stored.
* a granulocyte count of less than 1500/µl and a platelet count less than 150,000/µl.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2002-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Barlogie, MD, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences/MIRT, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Al Hadidi S, Ababneh OE, Schinke CD, Thanendrarajan S, Siegel ER, Bailey C, Smith R, Panozzo SB, Zangari M, Tricot G, Shaughnessy JD Jr, Zhan F, Sawyer J, Barlogie B, van Rhee F. Long-Term Follow-Up of Patients With Multiple Myeloma Treated on Earlier Total Therapy Protocols: A Secondary Analysis of 3 Clinical Trials. JAMA Oncol. 2025 Aug 1;11(8):910-915. doi: 10.1001/jamaoncol.2025.1394. PMID 40471585

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Treatment: Protocol therapy consists of a remission induction phase with mutually non-cross resistant combinations of vincristine, adriamycin, dexamethasone (VAD), high-dose cyclophosphamide with stem cell procurement and etoposide, dexamethasone, cytarabine, cisplatin (EDAP) followed by two courses of melphalan-based high-dose therapy supported by autologous stem cell transplants 4-6 months apart. Maintenance with interferon alpha will be administered until disease progression.
  VAD: 3 Cycles (3rd cycle optional):
  Vincristine 0.5 mg/d d 1 - 4 CI Adriamycin 10 mg/m2/d d 1 - 4 CI Dexamethasone 40 mg/d d 1-4, 9-12, 17-20
  High-Dose cyclophosphamide: Approximately 5-6 weeks after VAD 2 or 3:
  Cytoxan 1.2g/m2/d d 1 - 5 Mesna 3.6 g/m2 d 1
  Hemopoietic stem cell procurement: Collection target = 10 x 10^6 cells/kg
  EDAP: Approximately 5-6 weeks after high-dose cyclophosphamide
Period: Overall Study
Arm/Group | Study Treatment
Started | 231
Completed | 231
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Treatment
Number analyzed (Participants) | 231
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 211
  >=65 years | 20
Age, Continuous [Median (Full Range); unit: years] | 51.6 [26.5 to 71.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91
  Male | 140
Region of Enrollment [Number; unit: participants]
  United States | 231

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants That Are Relapse-free 5 Years After Initial Therapy
Description: Relapse is defined by the unequivocal objective evidence of recurrent disease such as:
  myeloma-related cytogenetic abnormalities; bone marrow plasmacytosis >10% or >5% light chain restricted, non-diploid, plasma cells on clg/DNA; new skeletal or MRI lesions; hypercalcemia not explained by any other cause; or reappearance of M-protein in blood or urine not related to immune recovery, recent infection, and present for >2 months.
Time Frame: 5 years
Measure: Number; unit: percentage of participants
Arm/Group | Study Treatment
Number analyzed (Participants) | 231
percentage of participants | 28

ADVERSE EVENTS:
Arm/Group | Study Treatment
Serious Adverse Events (participants affected / at risk) | 231/231
Other Adverse Events (participants affected / at risk) | 231/231
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Treatment (N=231)
Blood/bone marrow Grade 4 (Blood and lymphatic system disorders) | 155
Anemia Grade 4 (Blood and lymphatic system disorders) | 10
Neutropeni Grade 4 (Blood and lymphatic system disorders) | 136
WBC Grade 4 (Blood and lymphatic system disorders) | 150
Thrombocyt Grade 4 (Blood and lymphatic system disorders) | 37
Hepatobiliary/pancreas grade 3 (Endocrine disorders) | 41
Hepatobiliary/pancreas grade 4 (Endocrine disorders) | 1
Alkaline grade 3 (Endocrine disorders) | 5
Bilirubin grade 3 (Endocrine disorders) | 12
Bilirubin grade 4 (Endocrine disorders) | 1
Hypoalbumi grade 3 (Endocrine disorders) | 26
SGOT (AST) grade 3 (Endocrine disorders) | 4
SGPT (ALT) grade 3 (Endocrine disorders) | 8
Metabolic/laboratory grade 3 (Metabolism and nutrition disorders) | 89
Metabolic/laboratory grade 4 (Metabolism and nutrition disorders) | 28
Bicarbonat grade 3 (Metabolism and nutrition disorders) | 2
Hypercalce grade 3 (Metabolism and nutrition disorders) | 3
Hypercalce grade 4 (Metabolism and nutrition disorders) | 2
Hyperglyce grade 3 (Metabolism and nutrition disorders) | 15
Hyperglyce grade 4 (Metabolism and nutrition disorders) | 6
Hyperkalem grade 3 (Metabolism and nutrition disorders) | 7
Hyperkalem grade 4 (Metabolism and nutrition disorders) | 3
Hypermagne grade 3 (Metabolism and nutrition disorders) | 2
Hypematre grade 3 (Metabolism and nutrition disorders) | 2
Hypematre grade 4 (Metabolism and nutrition disorders) | 2
Hypocalcem grade 3 (Metabolism and nutrition disorders) | 11
Hypocalcem grade 4 (Metabolism and nutrition disorders) | 10
Hypokalemi grade 3 (Metabolism and nutrition disorders) | 39
Hypokalemi grade 4 (Metabolism and nutrition disorders) | 3
Hypomagnes grade 3 (Metabolism and nutrition disorders) | 4
Hypomagnes grade 4 (Metabolism and nutrition disorders) | 1
Hyponatrem grade 3 (Metabolism and nutrition disorders) | 34
Hyponatrem grade 4 (Metabolism and nutrition disorders) | 2
Hypophosph grade 3 (Metabolism and nutrition disorders) | 83
Hypophosph grade 4 (Metabolism and nutrition disorders) | 1
Renal/Genitourinary grade 3 (Renal and urinary disorders) | 14
Renal/Genitourinary grade 4 (Renal and urinary disorders) | 9
Creatinine grade 3 (Renal and urinary disorders) | 14
Creatinine grade 4 (Renal and urinary disorders) | 9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Study Treatment (N=231)
Anemia grade 2 (Blood and lymphatic system disorders) | 52
Thrombocyt grade 2 (Blood and lymphatic system disorders) | 34
Hepatobiliary/ pancreas grade 1 (Endocrine disorders) | 30
Hepatobiliary/pancreas grade 2 (Endocrine disorders) | 138
Alkaline grade 1 (Endocrine disorders) | 70
Alkaline grade 2 (Endocrine disorders) | 14
Bilirubin grade 1 (Endocrine disorders) | 38
Bilirubin grade 2 (Endocrine disorders) | 17
Hypoalbumi grade 1 (Endocrine disorders) | 34
Hypoalbumi grade 2 (Endocrine disorders) | 150
SGOT (AST) grade 1 (Endocrine disorders) | 78
SGOT (AST) grade 2 (Endocrine disorders) | 13
SGPT (ALT) grade 1 (Endocrine disorders) | 76
SGPT (ALT) grade 2 (Endocrine disorders) | 20
Metabolic/laboratory grade 2 (Metabolism and nutrition disorders) | 38
Bicarbonat grade 1 (Metabolism and nutrition disorders) | 97
Hypercalce grade 1 (Metabolism and nutrition disorders) | 17
Hyperglyce grade 1 (Metabolism and nutrition disorders) | 53
Hyperglyce grade 2 (Metabolism and nutrition disorders) | 55
Hyperkalem grade 1 (Metabolism and nutrition disorders) | 43
Hyperkalem grade 2 (Metabolism and nutrition disorders) | 29
Hypemagne grade 1 (Metabolism and nutrition disorders) | 27
Hypematre grade 1 (Metabolism and nutrition disorders) | 63
Hypocalcem grade 1 (Metabolism and nutrition disorders) | 71
Hypocalcem grade 2 (Metabolism and nutrition disorders) | 57
Hypokalemi grade 1 (Metabolism and nutrition disorders) | 105
Hypomagnes grade 1 (Metabolism and nutrition disorders) | 116
Hypomagnes grade 2 (Metabolism and nutrition disorders) | 25
Hyponatrem grade 1 (Metabolism and nutrition disorders) | 97
Hypophosph grade 2 (Metabolism and nutrition disorders) | 63
Renal/genitourinary grade 1 (Renal and urinary disorders) | 64
Renal/genitourinary grade 2 (Renal and urinary disorders) | 35
Creatinine grade 1 (Renal and urinary disorders) | 64
Creatinine grade 2 (Renal and urinary disorders) | 35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No